CLINICAL TRIAL: NCT00208247
Title: Cognitive-behavioural Therapy Versus Short-term Psychodynamic Psychotherapy: a Randomised Clinical Trial
Brief Title: KATHY:Cognitive-behavioural Therapy for Hypochondriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-11-DP-82-RKF-21
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Hypochondriasis
MeSH Terms: conditions — Hypochondriasis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- CBT (Experimental): The cognitive behavioural treatment developed by Salkovskis, Warwick and co-workers was used, with adaptations for the specific setting.
  Interventions: Behavioral: Cognitive behavioral psychotherapy
- STPP (Experimental): The short-term psychodynamic psychotherapy (STPP).
  Interventions: Behavioral: Cognitive behavioral psychotherapy
- Waiting List (Experimental): Patients in the waiting-list group were asked to keep in touch with their GP, who had been informed of the trial in writing. The patients and their GPs were instructed not to begin any other treatment during the study period. After 6 months, the patients on the waiting list were re-evaluated for inclusion and exclusion criteria and, if they still met the criteria, re-randomized to CBT or STPP.
  Interventions: Behavioral: Cognitive behavioral psychotherapy

INTERVENTIONS:
Behavioral: Cognitive behavioral psychotherapy

SUMMARY:
The purpose of this study was to examined if psychotherapy is an effecitive treatment for hypochondriasis.

DETAILED DESCRIPTION:
Background: The central feature of hypochondriasis is preoccupation or fear of having a serious disease based on misinterpretation of bodily signs. Psychotherapeutic treatments have developed with focus on different aspects of the condition. Several controlled trials have examined the effectiveness of different treatment strategies.

Hypothesis: Hypochondriasis is accessible for treatment. Specific cognitive treatment focused on misinterpretation of bodily sensations is more effective than short-term non-specific psychodynamic psychotherapy.

Method: Patients with hypochondriasis were randomisation to cognitive behavioural therapy (CBT), psychodynamic psychotherapy, or waiting list. Patients on waiting list were subsequently randomised to CBT or dynamic psychotherapy. The patients received six-teen sessions over a period of six month. Follow-up assessments were made six and twelve month after treatment.

ELIGIBILITY:
Inclusion Criteria:

(1) age between 18 and 65 years, (2) Danish as native language, (3) fulfilment of the ICD-10 research criteria for hypochondriasis (3), (4) health anxiety to a significant degree: a score more than 17 on the health anxiety inventory (HAI) (5).

-

Exclusion Criteria:

(1) current psychotic condition, (2) current substance abuse, (3) a medical condition which demanded immediate treatment, (4) psychopharmacological treatment initiated or increased during the last 6 weeks before treatment, and (5) previous cognitive behavioural treatment.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-12; Primary Completion 2003-01 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Two primary outcome measures were included 0, 6 and 12 month after treatment: the Health Anxiety Inventory (HAI), which is an 18-item, self-report questionnaire and the Hamilton Anxiety Rating Scale (HAM-A).

SECONDARY OUTCOMES:
Several secondary outcome measures were included 0, 6 and 12 month after treatment: Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Hamilton Rating Scale for Depression (HAM-D) and Global Assessment Functioning (GAF).

CONTACTS AND LOCATIONS:
Overall Officials: Morten Birket-Smith, DMSc, Study Director — Liaison Psychiatric Unit, Bispebjerg Hospital, 2400 NV Copenhagen, Denmark; Per Sorensen, MD, Principal Investigator — Liaison Psychiatric Unit, Bispebjerg Hospital, 2400-NV Copenhagen, Denmark